CLINICAL TRIAL: NCT03421015
Title: Genomic Analysis in Localized or Locally Advanced Prostate Cancer. Identification of Biomarkers Predictive of Biochemical or Metastatic Recurrence
Brief Title: Genetic Analysis of Prostate Cancer to Identify Predictive Markers of Disease Relapse or Metastatic Evolution
Acronym: CHRU-WCMC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Lille (Other)
Collaborators: Weill Medical College of Cornell University (Other); New York Presbyterian Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2017_12; 2017-A01870-53 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-01-29; First posted 2018-02-05 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Prostatic Neoplasms
Keywords: localized prostate cancer; prostatectomy; biomarkers; metastatic recurrence; genomic
MeSH Terms: conditions — Prostatic Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- case group: patients with biochemical recurrence and positive imaging (case group)
- Control Group: patients without biochemical recurrence (control group)

SUMMARY:
Developing a genetic study on localized or locally advanced prostate cancer. The aim of the study is to identify genomic alteration predictive of metastatic recurrence in the context of primary heterogeneity, by using the next generation sequencing (NGS) techniques.

Identifying such biomarkers may be useful to detect a higher relapse risk, and thus lower the mortality rate.

ELIGIBILITY:
Inclusion Criteria:

* Patients managed by radical prostatectomy for prostate cancer between 2000 and 2016.
* Follow up > 6 years
* Negative pre surgical extension assessment
* Prognostic Grade Groups (OGG) III-IV-V
* Biochemical recurrence defined by 2 consecutive PSA rises ≥ 0,2 ng/mL
* Metastasis positive imaging

Exclusion Criteria:

* Neoadjuvant therapy
* Follow up < 6 years
* Prognostic Grade Groups (PGG) I-II
* Biochemical recurrence with metastasis negative imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients managed by radical prostatectomy for prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
The genetic alteration frequencies of TMPRSS2-ERG gene fusion | Baseline

SECONDARY OUTCOMES:
Frequency of amplification of proto-oncogenes (MYC, AR, PIK3CA), | Baseline
Frequency of mutations or deletions of tumor suppressor genes (PTEN, TP53, NKX3-1), | Baseline
Frequency of point mutations modifying protein function (SPOP) | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Arnauld Villers, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Claude Huriez, CHRU, Lille, France